CLINICAL TRIAL: NCT06011785
Title: Using Silica 12CH to Mitigate the Effects and Symptoms of Silicosis in Brazil
Acronym: HOHM
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: HOHM Foundation (Other)
Responsible Party: Principal Investigator, Alastair Gray, Director Research, HOHM Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HOHMF
Record Dates: First submitted 2023-07-24; First posted 2023-08-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Silicosis
MeSH Terms: conditions — Silicosis | interventions — gp100 Melanoma Antigen

STUDY DESIGN:
Intervention Model Description: The study design is a controlled non-blinded clinical study without randomization to test the effectiveness of an intervention among individuals with symptoms of Silicosis as a result of working as quartzite miners. The intervention to be studied is a homeopathic preparation of Silica 12CH on a sample of clients with Silicosis already receiving ongoing conventional medical care. The intervention is Silica 12CH given over one year: a single dose at intervals of three months (three times in the study period).
  Participants will be recruited locally through the clinic where they already receive ongoing medical attention. The local secretary of health authorizes the release of the patient files. Potential participants will be given printed information about the study details along with information about how to participate and the associated deadlines for joining the study. Interested individuals will be given the informed consent form.
Masking Description: No masking required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental): Participants have Silicosis and wish to be included in the intervention group
  Interventions: Drug: Silica 12CH

INTERVENTIONS:
Drug: Silica 12CH — Participants will freely elect to be in either the intervention group. Individuals in the experimental group will receive the intervention while also following the standard-care protocol. All individuals will be encouraged to continue with any concurrent conventional medical treatment for their Silicosis-related symptoms. Individuals in either group may freely leave the study at any time with no consequence. Additionally, participants may freely elect to decide opt out at any time.
  Other Names: Silicea terra (sil)

SUMMARY:
This clinical study aims to address a research and clinical treatment gap related to individuals with symptoms of Silicosis resulting from quartzite mining work. Silicosis represents a challenge in this specific population in Sao Thome das Letras, Minas Gerais. Silicosis is a severe disease and is considered incurable. Current conventional medicine only offers palliative care for those with Silicosis, highlighting the important and urgent need for research into complementary care approaches.

DETAILED DESCRIPTION:
The study design is a simple clinical trial to assess the effect of the homeopathic medication Silica 12CH given alongside the conventional treatment of Silicosis, versus standard treatment alone for Silicosis.

The study design is a controlled non-blinded clinical study without randomization to test the effectiveness of a homeopathic intervention among individuals with symptoms of Silicosis as a result of working as quartzite miners. The intervention to be studied is a homeopathic preparation of Silica 12CH on a sample of clients with Silicosis already receiving ongoing conventional medical care. The intervention is Silica 12CH given over one year: a single dose at intervals of three months (three times in the study period).

Participants will be recruited locally through the clinic where they already receive ongoing medical attention. The local secretary of health authorizes the release of the patient files. Potential participants will be given printed information about the study details along with information about how to participate and the associated deadlines for joining the study. Interested individuals will be given the informed consent form.

Participants will freely elect to be in either the control or intervention group. Individuals in the control group follow the standard-care protocol without the homeopathic intervention. Individuals in the experimental group will receive the homeopathic intervention while also following the standard-care protocol. All individuals will be encouraged to continue with any concurrent conventional medical treatment for their Silicosis-related symptoms. Individuals in either group may freely leave the study at any time with no consequence. Additionally, participants may freely elect to be moved from the control group into the experimental group at the half-way point in the study.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate, participants must meet the following criteria:

  * must be at least 18 years old
  * must have a clinical diagnosis of silicosis
  * must be receiving conventional medical care and/or monitoring for their condition

Exclusion Criteria:

* ● Individuals under the age of 18

  * individuals who are not receiving conventional medical care and/or monitoring for their condition
  * individuals too infirm to receive regular monitoring as required for the study
  * Interested participants without Silicosis
  * Individuals with Tuberculosis
  * Individuals defined as part of a vulnerable group

    * legal or clinically incapable persons
    * person in a state of temporary disability;
    * of a member of indigenous community

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in pulmonary health of individuals with Silicosis as assessed by symptoms '1' and '2' using the Measure Yourself Concerns and Wellbeing (MYCaW validated) wellness measurement instrument. 0 = As good as it can be. 6 = As bad as it can be | One year
  Monitor changes using validated wellness measurement instrument

SECONDARY OUTCOMES:
Changes in pulmonary health of individuals with Silicosis as assessed by overall wellness scores using the Measure Yourself Concerns and Wellbeing (MYCaW validated) wellness measurement instrument. 0 = As good as it can be. 6 = As bad as it can be. | One year
  Monitor changes using validated wellness measurement instrument

CONTACTS AND LOCATIONS:
Overall Officials: Alastair C Gray, PhD, Principal Investigator — HOHM Foundation
Locations (1):
- HOHM Foundation, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Survey data will be collected and stored using Alchemer before being transferred to Excel. Only the Principal Investigators will have access to this data at the conclusion of the data collection portion of the study. This information will then be stored on a password protected secure file. It will not be printed or shared with anyone else for any purpose.
  The only research personnel who will have authority to use or have access to the information are the Principal (Alastair Gray) and Co-Investigator (Parker Pracjek).

REFERENCES:
- [Result] Souza TP, Watte G, Gusso AM, Souza R, Moreira JDS, Knorst MM. Silicosis prevalence and risk factors in semi-precious stone mining in Brazil. Am J Ind Med. 2017 Jun;60(6):529-536. doi: 10.1002/ajim.22719. PMID 28514023
- [Result] Souza TP, van Tongeren M, Monteiro I. Respiratory health and silicosis in artisanal mine workers in southern Brazil. Am J Ind Med. 2021 Jun;64(6):511-518. doi: 10.1002/ajim.23242. Epub 2021 Mar 28. PMID 33774816
- [Result] Carneiro AP, Braz NF, Algranti E, Bezerra OM, Araujo NP, Amaral Eng Hyg LS, Edme JL, Sobaszek A, Cherot-Kornobis N. Silica exposure and disease in semi-precious stone craftsmen, Minas Gerais, Brazil. Am J Ind Med. 2017 Mar;60(3):239-247. doi: 10.1002/ajim.22682. PMID 28195659
- [Result] Goyal KK. Two cases of pulmonary TB treated with homeopathy. Homeopathy. 2002 Jan;91(1):43-6. doi: 10.1054/homp.2001.0009. No abstract available. PMID 12371452
- [Result] Chand KS, Manchanda RK, Mittal R, Batra S, Banavaliker JN, De I. Homeopathic treatment in addition to standard care in multi drug resistant pulmonary tuberculosis: a randomized, double blind, placebo controlled clinical trial. Homeopathy. 2014 Apr;103(2):97-107. doi: 10.1016/j.homp.2013.12.003. PMID 24685414
- [Result] Hoeper MM, Welte T. Systemic inflammation, COPD, and pulmonary hypertension. Chest. 2007 Feb;131(2):634-5; author reply 635. doi: 10.1378/chest.06-2207. No abstract available. PMID 17296674
- [Result] Boccolini PMM, de Lima Sirio Boclin K, de Sousa IMC, Boccolini CS. Prevalence of complementary and alternative medicine use in Brazil: results of the National Health Survey, 2019. BMC Complement Med Ther. 2022 Aug 2;22(1):205. doi: 10.1186/s12906-022-03687-x. PMID 35918725